CLINICAL TRIAL: NCT01933217
Title: Efficacy of Methylphenidate for Management of Long-Term Attention Problems After Pediatric Traumatic Brain Injury (TBI)
Brief Title: Methylphenidate for Attention Problems After Pediatric TBI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1K23HD074683-01A1 (NIH)
Record Dates: First submitted 2013-07-15; First posted 2013-09-02 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-04

CONDITIONS: Traumatic Brain Injury; TBI; ADHD
Keywords: TBI; traumatic brain injury; ADHD; methylphenidate; Concerta; attention problems
MeSH Terms: conditions — Brain Injuries, Traumatic; Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methylphenidate (Experimental): The study medication will consist of identical capsules filled Concerta® over-encapsulated to preserve double-blinding. The weekly dosages will be low, medium, and high based on weight cut-offs. Participants weighing less than 25kg will receive 18mg (low), 27mg (medium), and 36mg (high) dosages and participants weighing above 25kg will receive 18mg (low), 36mg (medium), and 54mg (high) dosages during the 3-week upward titration trial. Weekly ratings monitoring behavioral and side effect symptoms score and the Pittsburgh Side Effects Rating Scale.
  Interventions: Drug: Methylphenidate
- Placebo (Placebo Comparator): The study medication will consist of identical capsules filled with an inert white power (placebo). Weekly ratings monitoring behavioral and side effect symptoms score and the Pittsburgh Side Effects Rating Scale.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate
  Other Names: Concerta
  Arms: Methylphenidate
Drug: Placebo
  Arms: Placebo

SUMMARY:
Traumatic Brain Injury (TBI) - methylphenidate treatment

DETAILED DESCRIPTION:
The objectives of the study are to (1) determine the efficacy and dose-response of methylphenidate treatment of attention problems after pediatric traumatic brain injury (TBI) and (2) provide a better understanding of the relationship of a prior history of attention deficit hyperactivity disorder (ADHD), ADHD subtypes after TBI, executive function, and attentional control to treatment efficacy. The proposed clinical trial will enroll 50 children, age 6-17 years, with attention problems >6 months after moderate to severe TBI into a randomized, double-blind, placebo-controlled, cross-over design trial with 3 dose conditions (low, medium, and high).

ELIGIBILITY:
Inclusion Criteria:

* Between ages of 6-17
* Sustained Moderate to Severe TBI
* TBI occurred at least 6 months prior to beginning the study
* TBI occurred no earlier than 5 years of age
* Positive endorsement of 6 out of 9 items on the Vanderbilt ADHD inattention or hyperactivity scale

Exclusion Criteria:

* History of developmental disability or mental retardation
* Current active participation in ADHD-related behavioral intervention
* History of psychiatric condition requiring an inpatient admission in past 12 months
* Actively taking medications with a contraindication to Concerta that cannot be discontinued
* Current use of stimulant medication or ADHD specific medications that cannot be discontinued
* Non-blunt head injury
* Family history of arrhythmia
* Pregnancy

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2013-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad Kurowski, MS, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Kurowski BG, Epstein JN, Pruitt DW, Horn PS, Altaye M, Wade SL. Benefits of Methylphenidate for Long-Term Attention Problems After Traumatic Brain Injury in Childhood: A Randomized, Double-Masked, Placebo-Controlled, Dose-Titration, Crossover Trial. J Head Trauma Rehabil. 2019 Mar/Apr;34(2):E1-E12. doi: 10.1097/HTR.0000000000000432. PMID 30169436

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period for the study was January 2014 through July 2017. Participants were recruited from a tertiary pediatric hospital in the Midwestern United States with a Level 1 trauma designation. 321 participants were screened for eligibility.
Pre-assignment Details: Of the 321 assessed for eligibility, 40 participants scheduled a baseline assessment. 163 did not meet inclusion criteria and 118 declined to participate. 26 of the 40 participants were enrolled and randomized. Of those not randomized, 5 dropped before baseline visit and 9 did not show for scheduled baseline visit.
Groups:
- Methylphenidate, Then Placebo: For the first week, participants received the low-dose Methylphenidate condition (Concerta® over-encapsulated). Over the subsequent 3 weeks, the dose was titrated based on medication response and side effects to determine the optimal dose used for week 4. At the end of week 4, participants crossed-over and repeated the same procedures for the placebo condition. No wash-out period was used.
  The weekly dosages were low, medium, and high based on weight cut-offs. Participants weighing less than 25kg will receive 18mg (low), 27mg (medium), and 36mg (high) dosages and participants weighing above 25kg will receive 18mg (low), 36mg (medium), and 54mg (high) dosages during the 3-week upward titration trial.
- Placebo, Then Methlyphenidate: For the first week, participants received the low-dose Placebo condition (white powder pills). Over the subsequent 3 weeks, the dose was titrated based on medication response and side effects to determine the optimal dose used for week 4. At the end of week 4, participants crossed-over and repeated the same procedures for the Methlyphenidate condition. No wash-out period was used.
  The weekly dosages were low, medium, and high based on weight cut-offs. Participants weighing less than 25kg will receive 18mg (low), 27mg (medium), and 36mg (high) dosages and participants weighing above 25kg will receive 18mg (low), 36mg (medium), and 54mg (high) dosages during the 3-week upward titration trial.
Period: Randomization (4 Weeks)
Arm/Group | Methylphenidate, Then Placebo | Placebo, Then Methlyphenidate
Started | 12 | 14
Completed | 10 | 10
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 1 | 1
Period: Crossover (4 Weeks)
Arm/Group | Methylphenidate, Then Placebo | Placebo, Then Methlyphenidate
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo, Then Methylphenidate: For the first week, participants received the low-dose Placebo condition (white powder pills). Over the subsequent 3 weeks, the dose was titrated based on medication response and side effects to determine the optimal dose used for week 4. At the end of week 4, participants crossed-over and repeated the same procedures for the Methlyphenidate condition. No wash-out period was used.
  The weekly dosages were low, medium, and high based on weight cut-offs. Participants weighing less than 25kg will receive 18mg (low), 27mg (medium), and 36mg (high) dosages and participants weighing above 25kg will receive 18mg (low), 36mg (medium), and 54mg (high) dosages during the 3-week upward titration trial.
- Total: Total of all reporting groups
Arm/Group | Methylphenidate, Then Placebo | Placebo, Then Methylphenidate | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 14 | 26
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Parent Outcome-Vanderbilt ADHD Parent Rating Scales (VADPRS)
Description: Changes in symptom ratings were assessed on the Vanderbilt ADHD parent rating scales (VADPRS). A measure of ADHD symptom severity (Total Symptom Score [TSS]) is computed by totaling the scores from items 1-18 (Inattentive +Hyperactive-impulse domains), with a rating of none=0, occasionally=1, often=2, very often=3, provided. Scores for inattentive and hyperactive-impulsive domains were generated by totaling the 9 symptoms in these domains, and a TSS was computed by totaling items across domains.
Time Frame: Reported at End of Methylphenidate Arm (Week 4 or 8)
Population: All participants who completed outcome data and full cross-over intervention
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Methylphenidate: For the first week, participants received the low-dose Methylphenidate condition (Concerta® over-encapsulated). Over the subsequent 3 weeks, the dose was titrated based on medication response and side effects to determine the optimal dose used for week 4.
  The weekly dosages were low, medium, and high based on weight cut-offs. Participants weighing less than 25kg will receive 18mg (low), 27mg (medium), and 36mg (high) dosages and participants weighing above 25kg will receive 18mg (low), 36mg (medium), and 54mg (high) dosages during the 3-week upward titration trial.
- Placebo: For the first week, participants received the low-dose Placebo condition (white powder pills). Over the subsequent 3 weeks, the dose was titrated based on medication response and side effects to determine the optimal dose used for week 4.
  The weekly dosages were low, medium, and high based on weight cut-offs. Participants weighing less than 25kg will receive 18mg (low), 27mg (medium), and 36mg (high) dosages and participants weighing above 25kg will receive 18mg (low), 36mg (medium), and 54mg (high) dosages during the 3-week upward titration trial.
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale
  Vanderbilt Parent TSS | 1.10 (.11) | 1.47 (.11)
  Vanderbilt Parent Hyperactive | .84 (.11) | 1.14 (.11)
  Vanderbilt Parent Inattentive | 1.37 (.12) | 1.79 (.12)

2. Primary Outcome: Parent Outcome-Behavior Rating Inventory of Executive Functioning (BRIEF)
Description: The Behavior Rating Inventory of Executive Functioning (BRIEF)-Parent was used to assess executive functioning behaviors. The global executive composite (GEC), behavior regulatory index (BRI), and metacognitive index (MI) T-scores were used, with higher scores reflecting poorer executive functioning. T-scores were normalized to 50 with a standard deviation of 10.
Time Frame: Reported at End of Methylphenidate Arm (Week 4 or 8)
Population: All participants who completed outcome data and full cross-over intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 20 | 20
score on a scale
  BRIEF GEC-Overall | 60.05 (1.30) | 65.20 (1.30)
  BRIEF BRI-Overall | 54.30 (1.33) | 58.00 (1.33)
  BRIEF MI-Overall | 62.40 (1.52) | 67.75 (1.52)

3. Secondary Outcome: Neuropsychological Outcome- Wechsler Intelligence Scale for Children, 4th Edition Processing Speed Index (WISC-IV-PSI)
Description: The Wechsler Intelligence Scale for Children, 4th Edition Processing Speed Index (WISC-IV-PSI) has been designed for children 6-16:11 years of age and provides a measure of processing speed. For this index scale, the average score is 100 with a standard deviation of 15. Higher scores reflect better processing speed. One participant was administered the Wechsler Adult Intelligence Scale 4th Edition Processing Speed Index (WAIS-IV-PSI). All scores were included in the combined WISC/WAIS processing speed variable since both measures yield highly correlated standard scores.
Time Frame: Reported at End of Methylphenidate Arm (Week 4 or 8)
Population: All participants who completed outcome data and full cross-over intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 20 | 20
score on a scale | 96.05 (2.24) | 91.25 (2.24)

4. Secondary Outcome: Teacher Outcome Measure
Description: Used to assess child behavior.
Time Frame: January 1, 2014 - July 20, 2017
Population: Challenges with engaging teachers made it difficult to collect teacher outcome measures.
Arm/Group | Methylphenidate, Then Placebo | Placebo, Then Methlyphenidate
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Weeks 1-8
Arm/Group | Methylphenidate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylphenidate (N=20) | Placebo (N=20)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No